CLINICAL TRIAL: NCT06374368
Title: Jejuno-Ileal and Jejuno-Colic Diversion as a New Bariatric Method in the Treatment of Diabetes and Obesity: Study Protocol for a Prospective Randomised Clinical Trial
Brief Title: Small Bowel Diversion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ostrava (Other)
Collaborators: Institute for Clinical and Experimental Medicine (Other Government); Vitkovice Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JID-SURG
Record Dates: First submitted 2021-12-02; First posted 2024-04-18 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Type2 Diabetes
Keywords: Obesity; Type 2 Diabetes; Partial Jejunal Diversion; Partial Jejuno-colic Diversion; Bariatric surgery; Metabolic surgery; Side-to-Side Anastomosis
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- obese patients with jejuno-ileal diversion (Active Comparator): Jejuno-ileal diversion without gastric restriction using standard bariatric surgical technique with standard staplers and surgical suturing.
  Interventions: Procedure: jejuno-ileal diversion
- obese patients with jejuno-colic diversion (Active Comparator): Jejuno-colic diversion without gastric restriction using standard bariatric surgical technique with standard staplers and surgical suturing
  Interventions: Procedure: jejuno-colic diversion

INTERVENTIONS:
Procedure: jejuno-ileal diversion — The surgery is performed in general anesthesia with orotracheal intubation. The laparoscopic approach is used. After establishing pneumoperitoneum (insufluation of the abdominal cavity with CO2) the 1th. trocar and laparoscopic camera are introduced through small incision. After visual control of abdominal cavity additional 2-3 trocars for operating instruments are introduced. The site of future anastomosis is identified (45 cm from ligament of Treitz on jejunum and 45 cm for the ileocoecal junction on ileum). The anastomosis between these two parts of jejunum and ileum is created by the means of linear stapler (45 mm).
  Arms: obese patients with jejuno-ileal diversion
Procedure: jejuno-colic diversion — The surgery is performed in general anesthesia with orotracheal intubation. The laparoscopic approach is used. After establishing pneumoperitoneum (insufluation of the abdominal cavity with CO2) the 1th. trocar and laparoscopic camera are introduced through small incision. After visual control of abdominal cavity additional 2-3 trocars for operating instruments are introduced. The anastomosis is created between jejunum (45 from ligament of Treitz) and transverse colon (behind the liver flexure).
  Arms: obese patients with jejuno-colic diversion

SUMMARY:
In an effort to replicate metabolic surgery's durable results in metabolic disease while minimizing its risks, two innovative methods has been created. Two surgical methods to create a bowel-to-bowel anastomosis, similar to the type used in current metabolic surgeries. It be to create a jejuno-ileal, side-to-side anastomosis and jejunocolic side-to-side anastomosis. The side-to-side jejuno-ileal anastomosis and side-to-side jejunocolic anastomosis provides two routes for ingested food. The new, shorter route has a malabsorptive effect similar to that seen in Roux en-Y gastric bypass (RYGB) and biliopancreatic diversion (BPD) - procedures which leads to weight loss. Additionally, delivery of non-absorbed macronutrients to the distal ileum, or transverse colon can enhance incretin effect and improve Type 2 Diabetes Mellitus parameters. However, the native route is also preserved, which theoretically reduces the risk of malnutrition, diarrhea, and metabolic derangements seen in other metabolic surgeries.The side-to-side jejuno-ileal anastomosis was already tested in the Pilot Study of the GI Windows Self-Forming Magnetic (SFM) Anastomosis Device for Creation of an Incisionless Small Bowel Bypass for Treatment of Obesity and Diabetes in year 2015 (15). The results of this study demonstrated the safety of this approach without serious adverse events. This non-surgical approach resulted in significant weight loss, favorable changes in insulin and incretin responses to a mixed meal and significant improvement in HbA1c in T2DM (16).In summary, metabolic diseases are a growing pandemic with suboptimal clinical solutions. The surgical side-to-side jejuno-ileal anastomosis and side-to-side jejuno-colic anastomosis without gastrectomy potentially represents a new class of therapy that may produce durable clinical results generally associated with surgery while minimizing its attendant risks.

DETAILED DESCRIPTION:
The study subjects who meet Inclusion criteria and baseline procedures undergo surgery (jejunal-ileal diversion/ jejuno-colic diversion). The surgery is performed in general anesthesia with orotracheal intubation. The laparoscopic approach is used. After establishing pneumoperitoneum (insufluation of the abdominal cavity with CO2) the 1th. trocar and laparoscopic camera are introduced through small incision. After visual control of abdominal cavity additional 2-3 trocars for operating instruments are introduced. The site of future anastomosis is identified (45 cm from ligament of Treitz on jejunum and 45 cm for the ileocoecal junction on ileum). The anastomosis between these two parts of jejunum and ileum is created by the means of linear stapler (45 mm), The residual defect is closed by manual continuous suture. The food will be passed through intestine partially through whole small intestine and partially through the anastomosis. In the second group of patients is the anastomosis created between jejunum (45 from ligament of Treitz) and transverse colon (behind the liver flexure) by means of the same technique. Before the end of the operation the control of bleeding is performed. Afterwards the trocars are removed under visual control. The pneumoperitoneum is released and the incisions are sutured. The subject will have follow-up clinic visits specific to the study at weeks 1, 2, and 3 and at months 1, 2, 3, 6, 12, 18, 24, 30 and 36 after the original procedure. At each clinic visit, the subject will undergo review of medical history, assessment for adverse events, physical examination (including weight and girth measurements) and blood work (e.g. glycated hemoglobin HbA1c). At specific intervals, principal metabolic studies will be performed, including a mixed meal tolerance test. Upper GI series radiographic studies at baseline and 14days after procedure as well as at the discretion of the principal investigator, will be performed, focusing on the patency of the anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years at screening;
* Body mass index ≥30 or ≤50kg/m2;
* If subject has Type 2 Diabetes: fasting plasma glucose greater than 6,1 mmol/l at time of enrollment if not treated with anti-diabetic medication;
* If on no diabetes medications, Hemoglobin A1C between and including 6.5 and 9.0 at time of enrollment.

Exclusion Criteria:

* Body Mass Index >50 or <30 kg/m2;
* Diagnosis of Type 2 diabetes less than 6 months;
* History of suspected gastrointestinal disease (for example cirrhosis, inflammatory bowel disease);
* History of active malignancy (not in remission) with the exception of squamous or basal cell carcinoma of the skin;
* Ongoing systemic infection;
* Chronic pancreatitis;
* Chronic liver disease of any cause;
* Poorly controlled psychiatric disease (for example ongoing major depression, schizophrenia, borderline personality, suicidality, psychosis);
* Any history of an eating disorder within the past 5 years;
* Pre-existing severe comorbid cardio-respiratory disease (for example congestive heart failure, cardiac arrhythmia, coronary artery disease, chronic obstructive lung disease, pulmonary embolism);
* uncontrolled hypertension (systolic Blood Preassure > 150 mm Hg or diastolic Blood Preassure > 100 mm Hg).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Total body weight loss | 36 months
  Weight change in percentage
Glycated hemoglobin loss | 36 months
  Glycated hemoglobin change in blood
Diabetes medication loss | 36 months
  Reduction in diabetes medication requirements (for diabetic cohort) - absolute value
Total cholesterol loss | 36 months
  Total cholesterol loss in blood
Low density lipoprotein loss | 36 months
  Low density lipoprotein loss in blood
High density lipoprotein loss | 36 months
  High density lipoprotein loss in blood
Leptin metabolism evaluation | 36 months
  Leptin value increase/decrease in blood
Adiponectin metabolism evaluation | 36 months
  Adiponectin value increase/decrease in blood
Bile acids metabolism evaluation | 36 months
  Bile acids value increase/decrease in blood

SECONDARY OUTCOMES:
Change from baseline quality of life-Lite | 36 months
  Questionary "Weight on Quality of Life-Lite (IWQOL-Lite)"
Change from baseline quality of life - Sort Form Survey | 36 months
  Questionary "36-Item Short Form Survey (SF-36)"

CONTACTS AND LOCATIONS:
Overall Officials: Marek Bužga, Doc., Principal Investigator — University of Ostrava
Locations (2):
- Czechia (2):
  - University of Ostrava, Ostrava
  - University of Ostrava, Faculty of Medicine, Ostrava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walpole SC, Prieto-Merino D, Edwards P, Cleland J, Stevens G, Roberts I. The weight of nations: an estimation of adult human biomass. BMC Public Health. 2012 Jun 18;12:439. doi: 10.1186/1471-2458-12-439. PMID 22709383
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Fried M, Yumuk V, Oppert JM, Scopinaro N, Torres AJ, Weiner R, Yashkov Y, Fruhbeck G; European Association for the Study of Obesity; International Federation for the Surgery of Obesity - European Chapter. Interdisciplinary European Guidelines on metabolic and bariatric surgery. Obes Facts. 2013;6(5):449-68. doi: 10.1159/000355480. Epub 2013 Oct 11. PMID 24135948
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Danaei G, Finucane MM, Lu Y, Singh GM, Cowan MJ, Paciorek CJ, Lin JK, Farzadfar F, Khang YH, Stevens GA, Rao M, Ali MK, Riley LM, Robinson CA, Ezzati M; Global Burden of Metabolic Risk Factors of Chronic Diseases Collaborating Group (Blood Glucose). National, regional, and global trends in fasting plasma glucose and diabetes prevalence since 1980: systematic analysis of health examination surveys and epidemiological studies with 370 country-years and 2.7 million participants. Lancet. 2011 Jul 2;378(9785):31-40. doi: 10.1016/S0140-6736(11)60679-X. Epub 2011 Jun 24. PMID 21705069
- [Background] Hofso D, Jenssen T, Hager H, Roislien J, Hjelmesaeth J. Fasting plasma glucose in the screening for type 2 diabetes in morbidly obese subjects. Obes Surg. 2010 Mar;20(3):302-7. doi: 10.1007/s11695-009-0022-5. Epub 2009 Dec 1. PMID 19949889
- [Background] Honzikova N, Krticka A, Zavodna E, Javorka M, Tonhajzerova I, Javorka K. Spectral peak frequency in low-frequency band in cross spectra of blood pressure and heart rate fluctuations in young type 1 diabetic patients. Physiol Res. 2012;61(4):347-54. doi: 10.33549/physiolres.932300. Epub 2012 Jun 6. PMID 22670692
- [Background] Rubino F, Nathan DM, Eckel RH, Schauer PR, Alberti KG, Zimmet PZ, Del Prato S, Ji L, Sadikot SM, Herman WH, Amiel SA, Kaplan LM, Taroncher-Oldenburg G, Cummings DE; Delegates of the 2nd Diabetes Surgery Summit. Metabolic Surgery in the Treatment Algorithm for Type 2 Diabetes: a Joint Statement by International Diabetes Organizations. Obes Surg. 2017 Jan;27(1):2-21. doi: 10.1007/s11695-016-2457-9. PMID 27957699
- [Background] Adams TD, Arterburn DE, Nathan DM, Eckel RH. Clinical Outcomes of Metabolic Surgery: Microvascular and Macrovascular Complications. Diabetes Care. 2016 Jun;39(6):912-23. doi: 10.2337/dc16-0157. PMID 27222549
- [Background] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Leccesi L, Nanni G, Pomp A, Castagneto M, Ghirlanda G, Rubino F. Bariatric surgery versus conventional medical therapy for type 2 diabetes. N Engl J Med. 2012 Apr 26;366(17):1577-85. doi: 10.1056/NEJMoa1200111. Epub 2012 Mar 26. PMID 22449317
- [Background] Rubino F, Gagner M. Potential of surgery for curing type 2 diabetes mellitus. Ann Surg. 2002 Nov;236(5):554-9. doi: 10.1097/00000658-200211000-00003. PMID 12409659
- [Background] Chang SH, Stoll CR, Song J, Varela JE, Eagon CJ, Colditz GA. The effectiveness and risks of bariatric surgery: an updated systematic review and meta-analysis, 2003-2012. JAMA Surg. 2014 Mar;149(3):275-87. doi: 10.1001/jamasurg.2013.3654. PMID 24352617
- [Background] Rubino F, Gagner M, Gentileschi P, Kini S, Fukuyama S, Feng J, Diamond E. The early effect of the Roux-en-Y gastric bypass on hormones involved in body weight regulation and glucose metabolism. Ann Surg. 2004 Aug;240(2):236-42. doi: 10.1097/01.sla.0000133117.12646.48. PMID 15273546
- [Background] Korner J, Inabnet W, Conwell IM, Taveras C, Daud A, Olivero-Rivera L, Restuccia NL, Bessler M. Differential effects of gastric bypass and banding on circulating gut hormone and leptin levels. Obesity (Silver Spring). 2006 Sep;14(9):1553-61. doi: 10.1038/oby.2006.179. PMID 17030966
- [Background] Laferrere B, Heshka S, Wang K, Khan Y, McGinty J, Teixeira J, Hart AB, Olivan B. Incretin levels and effect are markedly enhanced 1 month after Roux-en-Y gastric bypass surgery in obese patients with type 2 diabetes. Diabetes Care. 2007 Jul;30(7):1709-16. doi: 10.2337/dc06-1549. Epub 2007 Apr 6. PMID 17416796
- [Background] Rubino F, R'bibo SL, del Genio F, Mazumdar M, McGraw TE. Metabolic surgery: the role of the gastrointestinal tract in diabetes mellitus. Nat Rev Endocrinol. 2010 Feb;6(2):102-9. doi: 10.1038/nrendo.2009.268. PMID 20098450
- [Background] Ponnusamy V, Owens AP, Purkayastha S, Iodice V, Mathias CJ. Orthostatic intolerance and autonomic dysfunction following bariatric surgery: A retrospective study and review of the literature. Auton Neurosci. 2016 Jul;198:1-7. doi: 10.1016/j.autneu.2016.05.003. Epub 2016 May 31. PMID 27292926
- [Background] Straznicky NE, Eikelis N, Nestel PJ, Dixon JB, Dawood T, Grima MT, Sari CI, Schlaich MP, Esler MD, Tilbrook AJ, Lambert GW, Lambert EA. Baseline sympathetic nervous system activity predicts dietary weight loss in obese metabolic syndrome subjects. J Clin Endocrinol Metab. 2012 Feb;97(2):605-13. doi: 10.1210/jc.2011-2320. Epub 2011 Nov 16. PMID 22090279
- [Background] Casellini CM, Parson HK, Hodges K, Edwards JF, Lieb DC, Wohlgemuth SD, Vinik AI. Bariatric Surgery Restores Cardiac and Sudomotor Autonomic C-Fiber Dysfunction towards Normal in Obese Subjects with Type 2 Diabetes. PLoS One. 2016 May 3;11(5):e0154211. doi: 10.1371/journal.pone.0154211. eCollection 2016. PMID 27137224
- [Background] Cummings DE, Overduin J, Foster-Schubert KE, Carlson MJ. Role of the bypassed proximal intestine in the anti-diabetic effects of bariatric surgery. Surg Obes Relat Dis. 2007 Mar-Apr;3(2):109-15. doi: 10.1016/j.soard.2007.02.003. No abstract available. PMID 17386391
- [Background] Moo TA, Rubino F. Gastrointestinal surgery as treatment for type 2 diabetes. Curr Opin Endocrinol Diabetes Obes. 2008 Apr;15(2):153-8. doi: 10.1097/MED.0b013e3282f88a0a. PMID 18316951